CLINICAL TRIAL: NCT03664362
Title: Cumulative Victimization and Women's Health Risks: Development of an Intervention
Brief Title: The BSHAPE Intervention Program for Safety and Health of Survivors of Cumulative Trauma
Acronym: BSHAPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IRB00101882; K99HD082350 (NIH); R00HD082350 (NIH)
Record Dates: First submitted 2018-09-04; First posted 2018-09-10 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Violence; Cumulative Trauma; HIV Risk; Stress; Mental Health; Reproductive Health; Empowerment
MeSH Terms: conditions — Psychological Well-Being; Empowerment

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The BSHAPE Intervention (Experimental): Participants in the BSHAPE intervention attend a 9 sessions program post-assessments which is a combination of individualized and group-based sessions.
  Interventions: Behavioral: The BSHAPE Intervention
- Usual care or no treatment control (No Intervention): Participants in the control arm either are receiving no services or are engaged in usual care provided by community-based/health care organizations

INTERVENTIONS:
Behavioral: The BSHAPE Intervention — The BSHAPE intervention program key elements include strengths based assessments, individualized plans and support based on priorities and needs, motivational interviewing strategies, psychoeducation (education with skill building exercises), mindfulness activities, danger assessment, safety planning, behavioral activation and linkage to community resources
  Arms: The BSHAPE Intervention

SUMMARY:
The goal of the BSHAPE study is to test a trauma informed, culturally tailored, multicomponent program entitled BSHAPE (Being Safe, Healthy, And Positively Empowered) for immigrant survivors of cumulative trauma.

DETAILED DESCRIPTION:
The central hypothesis is that the BSHAPE intervention will promote immigrant women's safety and health (e.g..,improved mental health, reduced physiological impact of stress and health inequities (especially reproductive-sexual health and HIV)), thus leading to overall empowerment.

The study will:

1. Conduct a feasibility and acceptability evaluation of the BSHAPE intervention.
2. Test the BSHAPE intervention for large scale implementation in community-based clinics and programs serving immigrant women.

The impact of BSHAPE will be evaluated in comparison to usual care in promoting safety and health outcomes among immigrant women with cumulative trauma experiences at post-intervention and at 6 and 12 months follow up.

ELIGIBILITY:
Inclusion Criteria:

* 18-55 years of age
* Self-identify as a female
* Born in Africa or foreign born from African descent
* Must have a current or past abusive romantic relationship
* Must be a survivor of cumulative trauma
* Clinically significant symptoms of PTSD and/or depression
* At least one sexual HIV risk behavior

Exclusion Criteria:

* Less than 18 years of age or more than age 55
* Self-identify as a male
* Not African-born immigrant or born outside the US
* Is not a survivor of cumulative trauma
* Does not meet clinically significant criteria of PTSD and/or depression
* Does not report at least one sexual HIV risk behavior

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — If identify as biologically female or transgender female
Enrollment: 144 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2022-02-19 (Actual); Study Completion 2022-02-19 (Actual)

PRIMARY OUTCOMES:
Change in depressive symptoms | Through study completion, an average of 1 year (Assessment time points: Baseline, 3 months, 6 months, 12 months)
  The Patient Health Questionnaire (PHQ-9) is a 9 item measure to assess depression symptoms based on the diagnostic criteria for major depressive disorder in the Diagnostic and Statistical Manual (DSM-IV). Each of the 9 items scores from 0 (not at all) to 3 (nearly every day).
Change in symptoms of post-traumatic stress disorder (PTSD) | Through study completion, an average of 1 year (Assessment time points: Baseline, 3 months, 6 months, 12 months)
  Harvard Trauma Questionnaire (16 items) is used to measure symptoms of PTSD derived from the DSM-IIR/DSM-IV criteria for PTSD. The scale for each question includes four categories of response: "Not at all," "A little," "Quite a bit," "Extremely," rated 1 to 4, respectively
Change in perceived stress | Through study completion, an average of 1 year (Assessment time points: Baseline, 3 months, 6 months, 12 months)
  The Perceived stress scale is a 10 item self-report measure of stress. It is designed to assess how stressed one feels in the past month. Item responses are rated on a 5-point scale ranging from 0 (Never) to 4 (Very often). Higher scores indicate higher perceived stress. This scale is scored by summing the answers to all items, for a highest score of 40. Scores 0-13 indicate low stress, 14-26 is moderate stress and 27-40 is considered high stress.
Change in sexual risk behaviors | Through study completion, an average of 1 year (Assessment time points: Baseline, 3 months, 6 months, 12 months)]
  The Safe Sex Behavior Questionnaire is a 27-item self-report measure that describes sexual behaviors such as condom usage, sexual communication, and high-risk sexual behaviors. Item responses are rated on a 4-point scale ranging from 1 (Never) to 4 (Always). There are no subscales, and all items are summed to create a total score. Higher scores indicate engagement in safer sexual behaviors
Change in empowerment related to safety as assessed by the MOVERS scale | Through study completion, an average of 1 year (Assessment time points: Baseline, 3 months, 6 months, 12 months)
  The MOVERS is a 13 item scale that measures empowerment within the domain of safety. Participants respond to each item using a five-point scale from 1- "never true" to 5 - "always true". A maximum total of 65 and minimum of 13. Higher scores indicate higher level of empowerment related to safety.

SECONDARY OUTCOMES:
Change in overall empowerment as assessed by the Personal Progress Scale-Revised | Through study completion, an average of 1 year (Assessment time points: Baseline, 3 months, 6 months, 12 months)
  The Personal Progress Scale-Revised is a 28 item self-report measure of empowerment designed to assess multiple areas associated with empowerment such as positive self-evaluation, self-esteem, ability to regulate emotional distress, gender-role and cultural identity awareness, self-efficacy, self-care, problem-solving, assertiveness skills, and access to resources. Item responses are rated on a 7-point scale ranging from 1 (Almost Never) to 7 (Almost Always). A total maximum composite score of 196 and a minimum of 28. Higher scores indicate higher level of empowerment.
Change in self-efficacy related to coping with trauma as assessed by the Trauma Coping Self-Efficacy scale | Through study completion, an average of 1 year (Assessment time points: Baseline, 3 months, 6 months, 12 months)]
  The Trauma Coping Self-Efficacy scale is a 9-item self-report scale aimed at assessing the belief in one's ability to cope with trauma. Items are rated in a 7-point scale ranging from 1 (Not at all capable) to 7 (Totally capable). All items are averaged, for a high score of seven. Higher scores indicate greater trauma coping self-efficacy.
Change in self-efficacy for HIV/Sexually Transmitted Infection (STI) prevention as assessed by the Self-Efficacy for STI-HIV Scale | Through study completion, an average of 1 year (Assessment time points: Baseline, 3 months, 6 months, 12 months)
  The Self-Efficacy for STI-HIV Scale measures an individual's perceived ability to practice STD and HIV prevention strategies. The measure consists of 10 self-report items which are rated on a 5-point scale ranging from 1 (Not Sure) to 5 (Completely sure). All items are summed for a total score that can range from 10-50 with higher scores indicating higher self-efficacy.
Change in HIV knowledge using the HIV Knowledge Questionnaire | Through study completion, an average of 1 year (Assessment time points: Baseline, 3 months, 6 months, 12 months)
  The HIV Knowledge Questionnaire is a 18-item self report measure designed to measure ones understanding of HIV transmission and prevention. Items are scored in a true-false format where one point is awarded for a correct answer. Incorrect answers and "don't know" is scored as zero. Items are summed for a total possible score of 18. Higher scores indicate greater knowledge about how HIV is transmitted and how it can be prevented.
Change in Sexually Transmitted Disease (STD) knowledge using the STD Knowledge Questionnaire | Through study completion, an average of 1 year (Assessment time points: Baseline, 3 months, 6 months, 12 months)
  The STD Knowledge Questionnaire is a 27-item self-report measure designed to assess knowledge of transmission and prevention of common STDs such as Gonorrhea, Chlamydia, Hepatitis B, Human Papilloma Virus (HPV), and Genital Warts. Items are scored on a true-false scale where one point is awarded for each correct response. No points are given for incorrect responses or "Don't know". Items are summed to create a highest possible score of 27, with higher scores indicating high knowledge of how to prevent and transmit STDs.
Change in attitudes for stress management as assessed by the Inventory of Positive Psychological Attitudes | Through study completion, an average of 1 year (Assessment time points: Baseline, 3 months, 6 months, 12 months)
  The Inventory of Positive Psychological Attitudes measures attitudes in different domains that can act as buffers to prevent stress and stress-related disorders. The 15 items measuring confidence during stress is used which measures one's ability to handle difficult times will be used. Item responses are scored on a 7-point scale ranging from 1 to 7 with a maximum total of 105 and a minimum of 7. Higher scores indicate greater resiliency.
Change in utilization of healthcare services | Through study completion, an average of 1 year (Assessment time points: Baseline, 3 months, 6 months, 12 months)
  The Health Care Utilization measure was adapted from the Women's Health Care Experiences Survey. This measure was created as a self-report measure to capture women's use of different health care related services such as physical checkups, HIV screening, family planning services, abortion services, and other healthcare needs. For each different category of service, the measure asks if the service was used, where the service was received, if the service is available and why it was not used (if applicable). Each service is treated as a separate question, providing unique data; no scores are summed or averaged.
Change in severity and frequency of violence | Through study completion, an average of 1 year (Assessment time points: Baseline, 3 months, 6 months, 12 months)
  The adapted version of the revised Conflict Tactics Scale (CTS) will be used to measure change in exposure to violence. The items on the CTS-2 are scored using the severity-times-frequency weighted score, as recommended by Straus (2004).
Change in physiological stress responses | Assessment time points, Baseline, 3 months and 6 months
  Saliva samples are used to measure change in physiological stress response

CONTACTS AND LOCATIONS:
Overall Officials: Bushra Sabri, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will only be available to the research team members of the project
Time Frame: Data will only be available for the duration of the project and one year after completion
Access Criteria: The de-identified data will only be shared on a secure encrypted website that is managed by Johns Hopkins University

REFERENCES:
- [Derived] Sabri B, Perrin N, Hagos M. The being safe, health and positively empowered pilot randomized controlled trial: A digital multicomponent intervention for immigrant women with cumulative exposures to violence. Cultur Divers Ethnic Minor Psychol. 2025 Apr;31(2):271-284. doi: 10.1037/cdp0000635. Epub 2024 Feb 8. PMID 38330368
- [Derived] Sabri B, Vroegindewey A, Hagos M. Development, feasibility, acceptability and preliminary evaluation of the internet and mobile phone-based BSHAPE intervention for Immigrant survivors of cumulative trauma. Contemp Clin Trials. 2021 Nov;110:106591. doi: 10.1016/j.cct.2021.106591. Epub 2021 Oct 7. PMID 34626840